CLINICAL TRIAL: NCT03768726
Title: 26-WEEK OPEN-LABEL EXTENSION STUDY EVALUATING THE SAFETY AND TOLERABILITY OF FLEXIBLE DOSES OF ORAL ZIPRASIDONE IN CHILDREN AND ADOLESCENTS WITH BIPOLAR I DISORDER (MOST RECENT EPISODE MANIC)
Brief Title: Extension Study Evaluating The Safety And Tolerability Of Flexible Doses Of Oral Ziprasidone In Children And Adolescents With Bipolar I Disorder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pfizer has decided to perform the pre-specified final analysis at the current enrollment using a re-estimation of the sample size.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1281201
Record Dates: First submitted 2018-11-19; First posted 2018-12-07 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Intervention Model Description: Subjects would completed A1281198 will be transitioned under double blind conditions to 26 weeks of treatment with flexibly dosed opened label ziprasidone.
Masking Description: Subjects who participate in A1281198 will be transitioned under double blind conditions (during the first two weeks of the study) to 26 weeks of treatment with flexibly dosed opened label ziprasidone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ziprasidone (Experimental): All investigational products will be provided by Pfizer and will include oral ziprasidone capsules of 20, 40, 60, and 80 mg strength. Matching placebo capsules will also be supplied for the initial 1-14 day dose transition period. During the transition period all subjects will receive both active ziprasidone and placebo capsules. The placebo capsules are used to maintain the blind to the treatment assignment of the subjects in A1281198 . All medication will be packaged in childproof blister cards with columns for AM and for PM capsules. During the dose transition period (Weeks 1-2, Days 1-14), subjects will receive a study drug blister card for each week of transition dosing. Subjects weighing greater than 45 kg will receive 2 weeks of transition medication, while subjects weighing less than 45 kg will receive 1 week of transition medication.
  Interventions: Drug: Ziprasidone; Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone — All investigational products will be provided by Pfizer and will include oral ziprasidone capsules of 20, 40, 60, and 80 mg strength. Matching placebo capsules will also be supplied for the initial 1-14 day dose transition period. During the transition period all subjects will receive both active ziprasidone and placebo capsules. The placebo capsules are used to maintain the blind to the treatment assignment of the subjects in A1281198 . All medication will be packaged in childproof blister cards with columns for AM and for PM capsules. During the dose transition period (Weeks 1-2, Days 1-14), subjects will receive a study drug blister card for each week of transition dosing. Subjects weighing greater than 45 kg will receive 2 weeks of transition medication, while subjects weighing less than 45 kg will receive 1 week of transition medication.
Drug: Placebo — All investigational products will be provided by Pfizer and will include oral ziprasidone capsules of 20, 40, 60, and 80 mg strength. Matching placebo capsules will also be supplied for the initial 1-14 day dose transition period. During the transition period all subjects will receive both active ziprasidone and placebo capsules. The placebo capsules are used to maintain the blind to the treatment assignment of the subjects in A1281198 . All medication will be packaged in childproof blister cards with columns for AM and for PM capsules. During the dose transition period (Weeks 1-2, Days 1-14), subjects will receive a study drug blister card for each week of transition dosing. Subjects weighing greater than 45 kg will receive 2 weeks of transition medication, while subjects weighing less than 45 kg will receive 1 week of transition medication.

SUMMARY:
This 26-week open-label extension study is designed to provide information on the safety and tolerability of oral ziprasidone (20-80 mg BID (twice daily) with meals) during long-term administration in children and adolescents with Bipolar I Disorder (current or most recent episode manic).

DETAILED DESCRIPTION:
Study A1281201 is a 6 month, open label extension study of the ongoing double blind, randomized, placebo controlled study of ziprasidone in pediatric Bipolar Disorder (Study A1281198). Study A1281201 will enroll adolescents aged 10 to 17 years with Bipolar I Disorder who have participated in double blind Study A1281198. In order to be enrolled in this open label extension trial, subjects must have met the enrollment criteria for Study A1281198, and must meet the inclusion and exclusion criteria for Study A1281201 at the extension study Baseline visit (last visit in the double blind study).

The purpose of adding this extension study to the ongoing Geodon pediatric bipolar program is to obtain additional longer term safety data in children and adolescents with Bipolar I disorder treated with ziprasidone.

ELIGIBILITY:
Inclusion Criteria

* Evidence of personally signed and dated informed consent document by the legal representative and an assent document by the subject .
* Subjects and their legal guardians who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* The subjects must have received investigational product in Study A1281198 before entering this open label extension.
* In the investigator's opinion, the subject must be likely to benefit from antipsychotic therapy .
* All fertile male subjects and female subjects of childbearing potential who are sexually active and/or their legal guardians, as appropriate, must agree that a highly effective method of contraception

Exclusion Criteria

* Any subjects from the preceding double blind trail who experienced a serious adverse event which required study medication to be discontinued and the subject to be withdrawn from the study. Subjects who experienced cardiac arrhythmias, conduction abnormalities, or QTc prolongation (confirmed and persistent Fridericia's correction (QTcF) >480 msec or increase from baseline QTcF >60 msec) during the preceding study.
* Subjects requiring any medications not allowed by the Concomitant Medication Table 12 (see "Concomitant Treatment(s)").
* Subjects who require treatment with drugs that are known to consistently prolong the QT interval (see Concomitant Medication Table 12).
* Subjects who are judged by the investigator as being at imminent risk of suicide.
* Subjects living in the same home as another study participant or having the same caregiver during the same enrollment period (Such subjects can be enrolled in the study at different times but may not be in the study at the same time).
* Subjects should be excluded or a risk assessment should be done to verify that it is safe for the subject to participate in the trial if the subject's responses on the C SSRS or other information based on the investigator's judgment indicate:

  * Suicide ideation associated with actual intent and a method or plan such that a positive response ('Yes') is made on items 4 or 5 of the suicidal ideation subscale of the C SSRS; or
  * Any suicide behaviors such that a determination of 'yes' is made to any of the suicide behavior items of the C SSRS.
* Pregnant female subjects, breastfeeding female subjects.
* Participation in other studies other than the preceding Study.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (9):
  - Medical Research Group of Central Florida, Orange City, Florida
  - Inova Clinical Trials and Research Centre, Fayetteville, Georgia
  - Attalla Consultants, LLC dba Institute for Behavioral Medicine, Smyrna, Georgia
  - Finger Lakes Clinical Research, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - AIM Trials, LLC, Plano, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Eastside Therapeutic Resource Inc dba Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Atkinson S, Bachinsky M, Raiter Y, Abreu P, Ianos C, Chappell P, Findling RL. 26-Week Open-Label Extension Study Evaluating the Safety and Tolerability of Flexible Doses of Oral Ziprasidone in Children and Adolescents with Bipolar I Disorder (Most Recent Episode Manic). J Child Adolesc Psychopharmacol. 2022 Oct;32(8):453-458. doi: 10.1089/cap.2022.0030. PMID 36282771
- [Derived] Findling RL, Atkinson S, Bachinsky M, Raiter Y, Abreu P, Ianos C, Chappell P. Efficacy, Safety, and Tolerability of Flexibly Dosed Ziprasidone in Children and Adolescents with Mania in Bipolar I Disorder: A Randomized Placebo-Controlled Replication Study. J Child Adolesc Psychopharmacol. 2022 Apr;32(3):143-152. doi: 10.1089/cap.2021.0121. Epub 2022 Apr 7. PMID 35394365
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A1281201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who participated in study A1281198 (NCT02075047) and consented for treatment with open label ziprasidone were enrolled in the current study A1281201 (NCT03768726).
Groups:
- Ziprasidone in A1281198 and A1281201: Participants who were on ziprasidone in study A1281198, continued to receive the same dose of ziprasidone, under similar double-blind conditions for maximum up to Week 2. Participants with body weight greater than or equal to (>=) 45 kilogram (kg) had a target total daily dose range of 120-160 milligram per day (mg/day) given in 2 divided doses with food. Participants with body weight less than (<) 45 kg had a target total daily dose range of 60-80 mg/day given in 2 divided doses with food. Participants who did not tolerate a dose of 80 mg/day were allowed to have a dose reduction. The minimum permitted dose was 40 mg/day (20 mg twice a day) for all participants. Any participant if unable to tolerate the ziprasidone during Week 1 was discontinued from the study. Post Week 2 up to Week 26, dosing was open label and flexible. Participants had a follow-up Visit to trial site at 1 Week after last dose. Adverse events were collected up to 35 days after last dose of medication.
- Placebo in A1281198 Then Ziprasidone in A1281201: Participants who were on placebo in study A1281198, received ziprasidone, under similar double-blind conditions up to Week 2 (with body weight >45 kg) or Week 1 (with body weight <45 kg) and during the respective specified duration dose was titrated-up, to the appropriate weight-adjusted target dose per discretion of the investigator to maintain optimal efficacy and tolerability. Dosing of ziprasidone was identical to A1281198 study. Any participant if unable to tolerate the ziprasidone during Week 1 was discontinued from the study. Post Week 2 or Week 1 (as applicable) up to Week 26, dosing was open label and flexible. Participants had a follow-up Visit to trial site at 1 Week after last dose. Adverse events were collected up to 35 days after last dose of study medication.
Period: Treatment Phase
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Started | 10 | 13
Completed | 2 | 10
Not Completed | 8 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal By Parent/Guardian | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1
Period: Follow-Up
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Started | 8 (Participants were followed up after completion or discontinuation of treatment.) | 12 (Participants were followed up after completion or discontinuation of treatment.)
Received Treatment | 8 | 12
Completed | 2 | 9
Not Completed | 6 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal By Parent/Guardian | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who took at least 1 dose of study medication in this open-label extension study.
Groups:
- Ziprasidone in A1281198 and A1281201: Participants who were on ziprasidone in study A1281198, continued to receive the same dose of ziprasidone, under similar double-blind conditions for maximum up to Week 2. Participants with body weight >=45 kg had a target total daily dose range of 120-160 mg/day given in 2 divided doses with food. Participants with body weight <45 kg had a target total daily dose range of 60-80 mg/day given in 2 divided doses with food. Participants who did not tolerate a dose of 80 mg/day were allowed to have a dose reduction. The minimum permitted dose was 40 mg/day (20 mg twice a day) for all participants. Any participant if unable to tolerate the ziprasidone during Week 1 was discontinued from the study. Post Week 2 up to Week 26, dosing was open label and flexible. Participants had a follow-up Visit to trial site at 1 Week after last dose. Adverse events were collected up to 35 days after last dose of medication.
- Total: Total of all reporting groups
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201 | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (2.3) | 14.2 (2.0) | 14.1 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 13 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 10 | 18
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. AEs included both serious and all non-serious AEs.
Time Frame: A1281201: Day 1 up to 35 days after last dose of study medication (maximum up to 31 Weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
Participants
  AEs | 7 | 12
  SAEs | 0 | 1

2. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hemoglobin (Hg), hematocrit, erythrocytes: <0.8*lower limits of normal (LLN); platelets: <0.5*LLN>1.75*upper limits of normal (ULN); leukocytes (leu), glucose-fasting:<0.6*LLN>1.5*ULN; lymphocytes (lym), lym/leu, neutrophils (neu), neu/leu, protein, albumin, phosphate, free thyroxine, thyroid stimulating hormone: <0.8*LLN>1.2*ULN; basophils (bas), bas/leu, eosinophils (eos), eos/leu, monocytes(mon), mon/leu: >1.2*ULN; bilirubin (total, direct, indirect):>1.5*ULN; aspartate aminotransferase(AT), alanine AT, lactate dehydrogenase, alkaline phosphatase:>3.0*ULN; blood urea nitrogen, creatinine, cholesterol (total, LDL, HDL), triglycerides, Hg A1C: >1.3*ULN; sodium: <0.95*LLN>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate: <0.9*LLLN>1.1*ULN; prolactin: >1.1*ULN; creatine kinase: >2.0*ULN; urobilinogen: >=1; Urine-specific gravity: <1.003>1.030, pH: <4.5 >8, glucose, protein, bilirubin, nitrite, leukocyte esterase, ketones: >=1.
Time Frame: A1281201: Day 1 up to 1 Week after last dose of study medication (maximum up to 27 Weeks)
Population: The safety analysis set included all participants who took at least 1 dose of study medication in this open-label extension study. Here 'Overall Number of Participants Analyzed' signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 8 | 13
Participants | 5 | 11

3. Secondary Outcome: Number of Participants With Physical Examination Abnormalities at Baseline and Week 26
Description: Parameters assessed for physical examination included: oral/tympanic temperature, general appearance, skin, head, ears, eyes, nose, throat, heart, lungs, breasts (if medically indicated), abdomen, external genitalia (if medically indicated), extremities, back/spinal system, lymph nodes or worsening of medical history conditions. Abnormality in physical examination was at the investigator's discretion.
Time Frame: Baseline (last measurement from A1281198), Week 26 of A1281201
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
Participants
  Baseline | 0 | 0
  Week 26 | 0 | 0

4. Secondary Outcome: Change From Baseline in Blood Pressure at Week 1, 2, 4, 6, 10, 14, 18, 22, 26 and Follow-up Visit
Description: Change from baseline in sitting and standing systolic and diastolic blood pressure in millimeter of mercury (mmHg) was reported.
Time Frame: Baseline (last measurement from A1281198), A1281201: Week 1, 2, 4, 6, 10, 14, 18, 22, 26, and Follow-up Visit (1 Week from last dose of study medication, anytime maximum up to Week 27)
Population: The safety analysis set included all participants who took at least 1 dose of study medication in this open-label extension study. Here 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
mmHg
  Sitting Systolic Blood Pressure, Baseline | 111.70 (13.712) | 111.38 (11.384)
  Sitting Systolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 9 | 12
  Sitting Systolic Blood Pressure, Change at Week 1 | 2.44 (10.944) | -1.00 (11.505)
  Sitting Systolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 7 | 12
  Sitting Systolic Blood Pressure, Change at Week 2 | 0.43 (6.024) | 0.08 (10.431)
  Sitting Systolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 7 | 12
  Sitting Systolic Blood Pressure, Change at Week 4 | 3.29 (8.036) | -1.83 (8.321)
  Sitting Systolic Blood Pressure, Change at Week 6: number analyzed (Participants) | 6 | 11
  Sitting Systolic Blood Pressure, Change at Week 6 | 3.17 (6.969) | -3.45 (11.903)
  Sitting Systolic Blood Pressure, Change at Week 10: number analyzed (Participants) | 5 | 11
  Sitting Systolic Blood Pressure, Change at Week 10 | -0.80 (9.203) | -3.09 (11.674)
  Sitting Systolic Blood Pressure, Change at Week 14: number analyzed (Participants) | 5 | 11
  Sitting Systolic Blood Pressure, Change at Week 14 | -2.80 (9.011) | -7.09 (8.949)
  Sitting Systolic Blood Pressure, Change at Week 18: number analyzed (Participants) | 3 | 11
  Sitting Systolic Blood Pressure, Change at Week 18 | -2.67 (8.327) | -0.82 (10.852)
  Sitting Systolic Blood Pressure, Change at Week 22: number analyzed (Participants) | 2 | 10
  Sitting Systolic Blood Pressure, Change at Week 22 | -5.00 (1.414) | 1.40 (11.568)
  Sitting Systolic Blood Pressure, Change at Week 26: number analyzed (Participants) | 8 | 13
  Sitting Systolic Blood Pressure, Change at Week 26 | -0.63 (9.620) | -2.23 (14.219)
  Sitting Systolic Blood Pressure, Change at Follow up Visit: number analyzed (Participants) | 4 | 3
  Sitting Systolic Blood Pressure, Change at Follow up Visit | 0.75 (7.365) | 7.67 (4.041)
  Standing Systolic Blood Pressure, Baseline | 113.40 (10.690) | 111.38 (12.738)
  Standing Systolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 9 | 11
  Standing Systolic Blood Pressure, Change at Week 1 | -0.67 (11.916) | -1.00 (8.161)
  Standing Systolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 7 | 12
  Standing Systolic Blood Pressure, Change at Week 2 | 2.86 (13.753) | 1.33 (12.759)
  Standing Systolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 7 | 12
  Standing Systolic Blood Pressure, Change at Week 4 | -1.57 (7.138) | 2.17 (11.707)
  Standing Systolic Blood Pressure, Change at Week 6: number analyzed (Participants) | 6 | 11
  Standing Systolic Blood Pressure, Change at Week 6 | 1.67 (7.230) | -2.00 (14.457)
  Standing Systolic Blood Pressure, Change at Week 10: number analyzed (Participants) | 5 | 11
  Standing Systolic Blood Pressure, Change at Week 10 | -0.60 (9.423) | -2.18 (11.391)
  Standing Systolic Blood Pressure, Change at Week 14: number analyzed (Participants) | 5 | 11
  Standing Systolic Blood Pressure, Change at Week 14 | -0.80 (9.039) | -4.55 (6.933)
  Standing Systolic Blood Pressure, Change at Week 18: number analyzed (Participants) | 3 | 11
  Standing Systolic Blood Pressure, Change at Week 18 | -2.67 (8.327) | -1.73 (13.342)
  Standing Systolic Blood Pressure, Change at Week 22: number analyzed (Participants) | 2 | 10
  Standing Systolic Blood Pressure, Change at Week 22 | -7.00 (7.071) | 5.40 (13.006)
  Standing Systolic Blood Pressure, Change at Week 26: number analyzed (Participants) | 8 | 12
  Standing Systolic Blood Pressure, Change at Week 26 | -3.38 (7.230) | -5.33 (12.010)
  Standing Systolic Blood Pressure, Change at Follow up Visit: number analyzed (Participants) | 4 | 2
  Standing Systolic Blood Pressure, Change at Follow up Visit | -5.50 (8.544) | 2.50 (4.950)
  Sitting Diastolic Blood Pressure, Baseline | 71.00 (7.688) | 72.00 (9.256)
  Sitting Diastolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 9 | 12
  Sitting Diastolic Blood Pressure, Change at Week 1 | 0.67 (10.794) | -1.67 (9.633)
  Sitting Diastolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 7 | 12
  Sitting Diastolic Blood Pressure, Change at Week 2 | -4.14 (3.185) | 0.17 (8.376)
  Sitting Diastolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 7 | 12
  Sitting Diastolic Blood Pressure, Change at Week 4 | 0.14 (6.768) | -2.17 (10.744)
  Sitting Diastolic Blood Pressure, Change at Week 6: number analyzed (Participants) | 6 | 11
  Sitting Diastolic Blood Pressure, Change at Week 6 | -0.83 (8.183) | 1.00 (13.176)
  Sitting Diastolic Blood Pressure, Change at Week 10: number analyzed (Participants) | 5 | 11
  Sitting Diastolic Blood Pressure, Change at Week 10 | -3.40 (4.393) | -7.09 (10.387)
  Sitting Diastolic Blood Pressure, Change at Week 14: number analyzed (Participants) | 5 | 11
  Sitting Diastolic Blood Pressure, Change at Week 14 | -6.20 (6.058) | -3.91 (10.094)
  Sitting Diastolic Blood Pressure, Change at Week 18: number analyzed (Participants) | 3 | 11
  Sitting Diastolic Blood Pressure, Change at Week 18 | -2.67 (3.786) | 0.27 (15.186)
  Sitting Diastolic Blood Pressure, Change at Week 22: number analyzed (Participants) | 2 | 10
  Sitting Diastolic Blood Pressure, Change at Week 22 | -5.50 (2.121) | -1.30 (9.019)
  Sitting Diastolic Blood Pressure, Change at Week 26: number analyzed (Participants) | 8 | 13
  Sitting Diastolic Blood Pressure, Change at Week 26 | -2.50 (6.302) | -2.46 (10.548)
  Sitting Diastolic Blood Pressure, Change at Follow up Visit: number analyzed (Participants) | 4 | 3
  Sitting Diastolic Blood Pressure, Change at Follow up Visit | -1.75 (13.175) | -1.67 (8.145)
  Standing Diastolic Blood Pressure, Baseline | 73.90 (6.402) | 74.85 (4.930)
  Standing Diastolic Blood Pressure, Change at Week 1: number analyzed (Participants) | 9 | 11
  Standing Diastolic Blood Pressure, Change at Week 1 | -1.00 (7.483) | -4.45 (6.654)
  Standing Diastolic Blood Pressure, Change at Week 2: number analyzed (Participants) | 7 | 12
  Standing Diastolic Blood Pressure, Change at Week 2 | -4.14 (3.132) | -0.33 (4.924)
  Standing Diastolic Blood Pressure, Change at Week 4: number analyzed (Participants) | 7 | 12
  Standing Diastolic Blood Pressure, Change at Week 4 | -3.14 (7.625) | -2.67 (10.465)
  Standing Diastolic Blood Pressure, Change at Week 6: number analyzed (Participants) | 6 | 11
  Standing Diastolic Blood Pressure, Change at Week 6 | -1.17 (5.776) | -2.82 (7.910)
  Standing Diastolic Blood Pressure, Change at Week 10: number analyzed (Participants) | 5 | 11
  Standing Diastolic Blood Pressure, Change at Week 10 | 0.40 (5.941) | -4.36 (7.215)
  Standing Diastolic Blood Pressure, Change at Week 14: number analyzed (Participants) | 5 | 11
  Standing Diastolic Blood Pressure, Change at Week 14 | -3.00 (3.317) | -4.09 (7.516)
  Standing Diastolic Blood Pressure, Change at Week 18: number analyzed (Participants) | 3 | 11
  Standing Diastolic Blood Pressure, Change at Week 18 | -5.33 (3.055) | -0.91 (12.136)
  Standing Diastolic Blood Pressure, Change at Week 22: number analyzed (Participants) | 2 | 10
  Standing Diastolic Blood Pressure, Change at Week 22 | 0.00 (5.657) | -4.30 (10.646)
  Standing Diastolic Blood Pressure, Change at Week 26: number analyzed (Participants) | 8 | 12
  Standing Diastolic Blood Pressure, Change at Week 26 | -0.50 (4.408) | -4.33 (8.700)
  Standing Diastolic Blood Pressure, Change at Follow-up Visit: number analyzed (Participants) | 4 | 2
  Standing Diastolic Blood Pressure, Change at Follow-up Visit | -7.75 (10.905) | -3.00 (2.828)

5. Secondary Outcome: Change From Baseline in Pulse Rate at Week 1, 2, 4, 6, 10, 14, 18, 22, 26 and Follow-up Visit
Description: Change from baseline pulse rate in beats per minute was reported in sitting and standing positions.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
beats per minute
  Sitting, Baseline | 77.90 (9.678) | 73.38 (11.701)
  Sitting, Change at Week 1: number analyzed (Participants) | 9 | 12
  Sitting, Change at Week 1 | 0.78 (8.969) | 2.00 (9.254)
  Sitting, Change at Week 2: number analyzed (Participants) | 7 | 12
  Sitting, Change at Week 2 | 0.00 (6.758) | 8.08 (11.782)
  Sitting, Change at Week 4: number analyzed (Participants) | 7 | 12
  Sitting, Change at Week 4 | -3.29 (7.365) | 2.00 (9.789)
  Sitting, Change at Week 6: number analyzed (Participants) | 6 | 11
  Sitting, Change at Week 6 | -1.17 (7.139) | 2.00 (10.954)
  Sitting, Change at Week 10: number analyzed (Participants) | 5 | 11
  Sitting, Change at Week 10 | 3.40 (11.261) | 0.18 (14.098)
  Sitting, Change at Week 14: number analyzed (Participants) | 5 | 11
  Sitting, Change at Week 14 | -3.00 (14.799) | -0.91 (13.308)
  Sitting, Change at Week 18: number analyzed (Participants) | 3 | 11
  Sitting, Change at Week 18 | -0.33 (8.622) | 1.09 (10.606)
  Sitting, Change at Week 22: number analyzed (Participants) | 2 | 10
  Sitting, Change at Week 22 | -12.00 (8.485) | 4.30 (12.056)
  Sitting, Change at Week 26: number analyzed (Participants) | 8 | 13
  Sitting, Change at Week 26 | -2.50 (11.452) | -2.69 (8.5787)
  Sitting, Change at Follow-up Visit: number analyzed (Participants) | 4 | 3
  Sitting, Change at Follow-up Visit | -2.50 (9.469) | 2.67 (12.858)
  Standing, Baseline: number analyzed (Participants) | 9 | 12
  Standing, Baseline | 80.00 (11.303) | 83.08 (13.554)
  Standing, Change at Week 1: number analyzed (Participants) | 8 | 11
  Standing, Change at Week 1 | 2.75 (9.270) | 1.09 (11.709)
  Standing, Change at Week 2: number analyzed (Participants) | 6 | 11
  Standing, Change at Week 2 | 5.33 (7.528) | 7.18 (12.131)
  Standing, Change at Week 4: number analyzed (Participants) | 6 | 11
  Standing, Change at Week 4 | 2.67 (10.270) | 1.27 (17.641)
  Standing, Change at Week 6: number analyzed (Participants) | 5 | 10
  Standing, Change at Week 6 | -3.00 (6.000) | 0.70 (13.857)
  Standing, Change at Week 10: number analyzed (Participants) | 4 | 10
  Standing, Change at Week 10 | 6.00 (10.066) | -0.20 (12.017)
  Standing, Change at Week 14: number analyzed (Participants) | 5 | 10
  Standing, Change at Week 14 | -2.20 (13.236) | -6.00 (10.914)
  Standing, Change at Week 18: number analyzed (Participants) | 3 | 10
  Standing, Change at Week 18 | -2.00 (6.928) | 2.30 (13.639)
  Standing, Change at Week 22: number analyzed (Participants) | 2 | 10
  Standing, Change at Week 22 | -10.00 (2.828) | 2.50 (12.095)
  Standing, Change at Week 26: number analyzed (Participants) | 7 | 12
  Standing, Change at Week 26 | 2.86 (14.381) | -0.33 (10.680)
  Standing, Change at Follow-up Visit: number analyzed (Participants) | 3 | 2
  Standing, Change at Follow-up Visit | -3.33 (4.619) | -1.00 (21.213)

6. Secondary Outcome: Change From Baseline in Height and Waist Circumference at Week 6, 26 and Follow-up Visit
Description: Change from baseline in height and waist circumference in centimeter (cm) was reported.
Time Frame: Baseline (last measurement from A1281198), A1281201: Week 6, 26, and Follow-up Visit (1 Week from last dose of study medication, anytime maximum up to Week 27)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
cm
  Height, Baseline | 159.82 (10.182) | 161.69 (11.996)
  Height, Change at Week 6: number analyzed (Participants) | 6 | 11
  Height, Change at Week 6 | 0.27 (0.455) | 0.77 (0.984)
  Height, Change at Week 26: number analyzed (Participants) | 7 | 13
  Height, Change at Week 26 | 2.04 (1.938) | 0.55 (1.535)
  Height, Change at Follow-up Visit: number analyzed (Participants) | 3 | 3
  Height, Change at Follow-up Visit | 0.90 (1.562) | 2.42 (1.413)
  Waist Circumference, Baseline | 78.89 (11.278) | 80.23 (13.981)
  Waist Circumference, Change at Week 6: number analyzed (Participants) | 6 | 11
  Waist Circumference, Change at Week 6 | -0.94 (2.483) | 2.23 (7.527)
  Waist Circumference, Change at Week 26: number analyzed (Participants) | 7 | 13
  Waist Circumference, Change at Week 26 | -1.02 (2.278) | 1.29 (4.210)
  Waist Circumference, Change at Follow-up Visit: number analyzed (Participants) | 3 | 3
  Waist Circumference, Change at Follow-up Visit | -6.40 (13.777) | 2.01 (3.778)

7. Secondary Outcome: Change From Baseline in Body Weight at Week 6, 26 and Follow-up Visit
Description: Change from baseline in body weight in kilogram (kg) was reported.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
kg
  Baseline | 57.76 (17.634) | 62.40 (19.375)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.82 (1.343) | 0.78 (2.530)
  Change at Week 26: number analyzed (Participants) | 7 | 13
  Change at Week 26 | 1.62 (2.528) | 2.33 (4.431)
  Change at Follow-up Visit: number analyzed (Participants) | 3 | 3
  Change at Follow-up Visit | 1.47 (1.629) | 4.68 (2.639)

8. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 6, 26 and Follow-up Visit
Description: Change from baseline in BMI in kilogram per meter square (kg/m^2) was reported.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
kg/m^2
  Baseline | 22.31 (5.081) | 23.37 (4.709)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.38 (0.519) | 0.91 (2.234)
  Change at Week 26: number analyzed (Participants) | 7 | 13
  Change at Week 26 | 0.19 (0.954) | 0.78 (1.800)
  Change at Follow-up Visit: number analyzed (Participants) | 3 | 3
  Change at Follow-up Visit | 0.35 (0.589) | 1.54 (1.447)

9. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) Z-score at Week 6, 26 and Follow-up Visit
Description: BMI z-score was reported using the Children's Hospital of Philadelphia z-score calculator. Z-score is a statistical measure to describe whether a mean was above or below the standard. A z-score of 0 is equal to the mean and is considered normal. Lower numbers indicate values lower than the mean and higher numbers indicate values higher than the mean. Higher values are indicative of higher BMI.
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
z-score
  Baseline | 0.58 (1.187) | 1.06 (0.852)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.12 (0.122) | -0.02 (0.511)
  Change at Week 26: number analyzed (Participants) | 7 | 13
  Change at Week 26 | 0.21 (0.747) | 0.11 (0.506)
  Change at Follow-up Visit: number analyzed (Participants) | 3 | 3
  Change at Follow-up Visit | 0.01 (0.207) | 0.26 (0.330)

10. Secondary Outcome: Change From Baseline in Heart Rate at Day 1, Week 1, 2, 4, 6, 14, 22, 26 and Follow-up Visit
Description: Change from baseline in heart rate in beats per minute was reported.
Time Frame: Baseline of A1281198, Day 1 (last measurement from A1281198), A1281201: Week 1, 2, 4, 6, 14, 22, 26, and Follow-up Visit (1 Week from last dose of study medication, anytime maximum up to Week 27)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
beats per minute
  Baseline | 77.8 (9.19) | 71.5 (14.12)
  Change at Day 1: number analyzed (Participants) | 8 | 12
  Change at Day 1 | -4.0 (9.40) | -1.2 (9.09)
  Change at Week 1: number analyzed (Participants) | 9 | 12
  Change at Week 1 | -2.0 (19.24) | 0.4 (16.12)
  Change at Week 2: number analyzed (Participants) | 7 | 12
  Change at Week 2 | 7.4 (16.69) | 5.0 (16.28)
  Change at Week 4: number analyzed (Participants) | 7 | 12
  Change at Week 4 | -7.3 (8.08) | 0.4 (13.20)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | -5.0 (13.04) | -3.9 (14.49)
  Change at Week 14: number analyzed (Participants) | 5 | 11
  Change at Week 14 | -0.6 (15.22) | -2.6 (15.23)
  Change at Week 22: number analyzed (Participants) | 2 | 10
  Change at Week 22 | -5.0 (0.00) | 0.3 (16.99)
  Change at Week 26: number analyzed (Participants) | 8 | 13
  Change at Week 26 | -7.8 (12.33) | -3.0 (8.69)
  Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  Change at Follow-up Visit | -15.0 | -13.0

11. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters at Day 1, Week 1, 2, 4, 6, 14, 22, 26 and Follow-up Visit
Description: Change from baseline in PR interval, QT interval corrected using the Bazett's correction (QTcB), QT interval corrected using the Fridericia's formula (QTcF), QT interval, RR interval, QRS duration in millisecond (msec) was reported.
Time Frame: as for outcome 10
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
msec
  PR interval, Baseline | 145.3 (14.77) | 148.5 (14.47)
  PR interval, Change at Day 1: number analyzed (Participants) | 8 | 12
  PR interval, Change at Day 1 | 1.0 (9.07) | 0.4 (10.25)
  PR interval, Change at Week 1: number analyzed (Participants) | 9 | 12
  PR interval, Change at Week 1 | 3.6 (14.17) | -2.6 (9.17)
  PR interval, Change at Week 2: number analyzed (Participants) | 7 | 12
  PR interval, Change at Week 2 | -4.6 (9.22) | 2.3 (11.69)
  PR interval, Change at Week 4: number analyzed (Participants) | 7 | 12
  PR interval, Change at Week 4 | 3.0 (5.16) | 1.1 (10.17)
  PR interval, Change at Week 6: number analyzed (Participants) | 6 | 11
  PR interval, Change at Week 6 | 0.0 (12.60) | 4.0 (10.89)
  PR interval, Change at Week 14: number analyzed (Participants) | 5 | 11
  PR interval, Change at Week 14 | -6.8 (4.87) | -2.0 (9.42)
  PR interval, Change at Week 22: number analyzed (Participants) | 2 | 10
  PR interval, Change at Week 22 | 12.5 (17.68) | 1.7 (9.25)
  PR interval, Change at Week 26: number analyzed (Participants) | 8 | 13
  PR interval, Change at Week 26 | -0.3 (7.76) | -0.9 (12.70)
  PR interval, Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  PR interval, Change at Follow-up Visit | -3.0 | 17.0
  QTcB interval, Baseline | 415.8 (16.13) | 412.4 (18.87)
  QTcB interval, Change at Day 1: number analyzed (Participants) | 8 | 12
  QTcB interval, Change at Day 1 | 1.0 (13.31) | 2.2 (15.72)
  QTcB interval, Change at Week 1: number analyzed (Participants) | 9 | 12
  QTcB interval, Change at Week 1 | 1.2 (18.34) | 15.6 (21.74)
  QTcB interval, Change at Week 2: number analyzed (Participants) | 7 | 12
  QTcB interval, Change at Week 2 | 6.4 (17.58) | 11.4 (24.01)
  QTcB interval, Change at Week 4: number analyzed (Participants) | 7 | 12
  QTcB interval, Change at Week 4 | -7.4 (9.36) | 2.9 (18.81)
  QTcB interval, Change at Week 6: number analyzed (Participants) | 6 | 11
  QTcB interval, Change at Week 6 | 9.0 (23.04) | 0.2 (27.75)
  QTcB interval, Change at Week 14: number analyzed (Participants) | 5 | 11
  QTcB interval, Change at Week 14 | -5.0 (21.30) | 3.9 (24.20)
  QTcB interval, Change at Week 22: number analyzed (Participants) | 2 | 10
  QTcB interval, Change at Week 22 | 19.0 (8.49) | 8.9 (30.94)
  QTcB interval, Change at Week 26: number analyzed (Participants) | 8 | 13
  QTcB interval, Change at Week 26 | 3.0 (26.88) | 2.5 (21.43)
  QTcB interval, Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  QTcB interval, Change at Follow-up Visit | -14.0 | -5.0
  QTcF interval, Baseline | 398.5 (14.80) | 401.8 (18.57)
  QTcF interval, Change at Day 1: number analyzed (Participants) | 8 | 12
  QTcF interval, Change at Day 1 | 3.8 (13.36) | 2.3 (11.40)
  QTcF interval, Change at Week 1: number analyzed (Participants) | 9 | 12
  QTcF interval, Change at Week 1 | 3.0 (12.65) | 14.0 (13.74)
  QTcF interval, Change at Week 2: number analyzed (Participants) | 7 | 12
  QTcF interval, Change at Week 2 | -0.3 (15.30) | 5.8 (13.98)
  QTcF interval, Change at Week 4: number analyzed (Participants) | 7 | 12
  QTcF interval, Change at Week 4 | -1.3 (13.90) | 1.3 (12.87)
  QTcF interval, Change at Week 6: number analyzed (Participants) | 6 | 11
  QTcF interval, Change at Week 6 | 12.5 (17.21) | 3.2 (18.94)
  QTcF interval, Change at Week 14: number analyzed (Participants) | 5 | 11
  QTcF interval, Change at Week 14 | -4.6 (10.01) | 6.2 (12.62)
  QTcF interval, Change at Week 22: number analyzed (Participants) | 2 | 10
  QTcF interval, Change at Week 22 | 23.5 (7.78) | 7.0 (21.21)
  QTcF interval, Change at Week 26: number analyzed (Participants) | 8 | 13
  QTcF interval, Change at Week 26 | 10.6 (16.77) | 4.3 (17.51)
  QTcF interval, Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  QTcF interval, Change at Follow-up Visit | 0.0 | 6.0
  QT interval, Baseline | 366.3 (21.79) | 382.8 (35.86)
  QT interval, Change at Day 1: number analyzed (Participants) | 8 | 12
  QT interval, Change at Day 1 | 9.6 (22.88) | 2.2 (17.17)
  QT interval, Change at Week 1: number analyzed (Participants) | 9 | 12
  QT interval, Change at Week 1 | 7.8 (37.06) | 10.8 (29.55)
  QT interval, Change at Week 2: number analyzed (Participants) | 7 | 12
  QT interval, Change at Week 2 | -11.4 (32.93) | -4.1 (26.25)
  QT interval, Change at Week 4: number analyzed (Participants) | 7 | 12
  QT interval, Change at Week 4 | 10.4 (25.34) | -2.1 (25.98)
  QT interval, Change at Week 6: number analyzed (Participants) | 6 | 11
  QT interval, Change at Week 6 | 20.5 (26.71) | 9.0 (25.65)
  QT interval, Change at Week 14: number analyzed (Participants) | 5 | 11
  QT interval, Change at Week 14 | -3.4 (20.70) | 10.6 (21.47)
  QT interval, Change at Week 22: number analyzed (Participants) | 2 | 10
  QT interval, Change at Week 22 | 34.0 (5.66) | 4.1 (31.27)
  QT interval, Change at Week 26: number analyzed (Participants) | 8 | 13
  QT interval, Change at Week 26 | 24.5 (18.90) | 7.2 (20.99)
  QT interval, Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  QT interval, Change at Follow-up Visit | 23.0 | 26.0
  RR interval, Baseline | 781.0 (95.07) | 873.6 (171.26)
  RR interval, Change at Day 1: number analyzed (Participants) | 8 | 12
  RR interval, Change at Day 1 | 33.6 (100.49) | -5.7 (102.47)
  RR interval, Change at Week 1: number analyzed (Participants) | 9 | 12
  RR interval, Change at Week 1 | 30.7 (203.15) | -17.7 (187.46)
  RR interval, Change at Week 2: number analyzed (Participants) | 7 | 12
  RR interval, Change at Week 2 | -73.3 (161.14) | -61.2 (179.08)
  RR interval , Change at Week 4: number analyzed (Participants) | 7 | 12
  RR interval , Change at Week 4 | 70.1 (86.24) | -26.9 (159.35)
  RR interval, Change at Week 6: number analyzed (Participants) | 6 | 11
  RR interval, Change at Week 6 | 56.5 (152.31) | 40.6 (173.34)
  RR interval, Change at Week 14: number analyzed (Participants) | 5 | 11
  RR interval, Change at Week 14 | 3.6 (157.07) | 33.2 (169.68)
  RR interval, Change at Week 22: number analyzed (Participants) | 2 | 10
  RR interval, Change at Week 22 | 69.0 (12.73) | -13.7 (208.06)
  RR interval, Change at Week 26: number analyzed (Participants) | 8 | 13
  RR interval, Change at Week 26 | 99.1 (165.02) | 20.4 (111.79)
  RR interval, Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  RR interval, Change at Follow-up Visit | 134.0 | 134.0
  QRS duration, Baseline | 84.4 (7.23) | 85.8 (5.90)
  QRS duration, Change at Day 1: number analyzed (Participants) | 8 | 12
  QRS duration, Change at Day 1 | 2.1 (3.76) | 2.8 (3.41)
  QRS duration, Change at Week 1: number analyzed (Participants) | 9 | 12
  QRS duration, Change at Week 1 | 1.0 (3.54) | 3.8 (5.64)
  QRS duration, Change at Week 2: number analyzed (Participants) | 7 | 12
  QRS duration, Change at Week 2 | 0.1 (3.24) | 1.7 (6.31)
  QRS duration, Change at Week 4: number analyzed (Participants) | 7 | 12
  QRS duration, Change at Week 4 | 2.0 (4.16) | 1.5 (5.25)
  QRS duration, Change at Week 6: number analyzed (Participants) | 6 | 11
  QRS duration, Change at Week 6 | -0.8 (3.06) | 2.5 (5.05)
  QRS duration, Change at Week 14: number analyzed (Participants) | 5 | 11
  QRS duration, Change at Week 14 | -1.2 (4.15) | 2.9 (7.30)
  QRS duration, Change at Week 22: number analyzed (Participants) | 2 | 10
  QRS duration, Change at Week 22 | 1.0 (2.83) | -0.3 (6.60)
  QRS duration, Change at Week 26: number analyzed (Participants) | 8 | 13
  QRS duration, Change at Week 26 | 3.5 (4.54) | 3.5 (4.93)
  QRS duration, Change at Follow-up Visit: number analyzed (Participants) | 1 | 1
  QRS duration, Change at Follow-up Visit | -4.0 | 11.0

12. Secondary Outcome: Change From Baseline in Simpson-Angus Rating Scale (SARS) Total Score at Week 1, 2, 4, 6, 10, 14, 18, 22, 26 and Follow-up Visit
Description: SARS: 10-item clinician rated instrument to assess parkinsonian symptoms and related extrapyramidal side effects. All 10 items were anchored on a 5-point scale: range 0 (absence of condition, normal) to 4 (the most extreme form of condition). Total score is sum of individual item scores, ranged from 0 (normal) to 40 (most extreme symptoms and effects); higher score indicates more affected. Rows with only non-zero data/values for change in SARS total score at specified time points, for at least 1 reporting arm, are reported below.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Baseline | 0.4 (1.26) | 0.0 (0.00)
  Change at Week 1: number analyzed (Participants) | 9 | 12
  Change at Week 1 | -0.2 (0.67) | 0.0 (0.00)
  Change at Week 2: number analyzed (Participants) | 7 | 12
  Change at Week 2 | 0.0 (0.00) | 0.2 (0.39)
  Change at Week 4: number analyzed (Participants) | 7 | 12
  Change at Week 4 | 0.0 (0.00) | 0.2 (0.58)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.0 (0.00) | 0.2 (0.40)
  Change at Week 26: number analyzed (Participants) | 8 | 13
  Change at Week 26 | -0.5 (1.41) | 0.0 (0.00)

13. Secondary Outcome: Change From Baseline in Global Clinical Assessment of Akathisia Subscale Score of Barnes Akathisia Rating Scale (BAS) at Week 1, 2, 4, 6, 10, 14, 18, 22, 26 and Follow-up Visit
Description: BAS: clinician rated scale to assess akathisia by determining the degree of subjective restlessness and distress associated with restlessness. Global clinical assessment of akathisia subscale score of BAS, was rated on a 6-point scale range 0 (no symptoms) to 5 (maximum severity of symptoms); higher score indicates increased severity.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Baseline | 0.0 (0.00) | 0.2 (0.38)
  Change at Week 1: number analyzed (Participants) | 9 | 12
  Change at Week 1 | 0.0 (0.00) | -0.1 (0.29)
  Change at Week 2: number analyzed (Participants) | 7 | 12
  Change at Week 2 | 0.0 (0.00) | 0.3 (1.07)
  Change at Week 4: number analyzed (Participants) | 7 | 12
  Change at Week 4 | 0.0 (0.00) | 0.1 (0.29)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.0 (0.00) | -0.2 (0.40)
  Change at Week 10: number analyzed (Participants) | 5 | 11
  Change at Week 10 | 0.0 (0.00) | -0.2 (0.40)
  Change at Week 14: number analyzed (Participants) | 5 | 11
  Change at Week 14 | 0.0 (0.00) | -0.2 (0.40)
  Change at Week 18: number analyzed (Participants) | 3 | 11
  Change at Week 18 | 0.0 (0.00) | -0.2 (0.40)
  Change at Week 22: number analyzed (Participants) | 2 | 10
  Change at Week 22 | 0.0 (0.00) | -0.2 (0.42)
  Change at Week 26: number analyzed (Participants) | 8 | 13
  Change at Week 26 | 0.0 (0.00) | -0.2 (0.38)
  Change at Follow-up Visit: number analyzed (Participants) | 2 | 3
  Change at Follow-up Visit | 0.0 (0.00) | -0.3 (0.58)

14. Secondary Outcome: Change From Baseline in Movement Cluster Subscale Score of Abnormal Involuntary Movement Scale (AIMS) at Week 1, 2, 4, 6, 10, 14, 18, 22, 26 and Follow-up Visit
Description: AIMS: clinician rated 12-item scale to document occurrences of dyskinesia in participants, specifically tardive dyskinesia. Items 1 to 10, scored as 0 (none) to 4 (severe); higher score indicates greater severity. Items 11 to 12 are questions with No or Yes response. Only the sum of the first 7 items were calculated to evaluate AIMS movement cluster subscale score, giving it a possible score range of 0 (none) to 28 (maximum severity), higher scores indicate greater severity. Rows with only non-zero data/values for change in AIMS-movement cluster subscale score at specified time points, for at least 1 reporting arm, are reported below.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Change at Week 2: number analyzed (Participants) | 7 | 12
  Change at Week 2 | 0.0 (0.00) | 0.3 (0.87)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.0 (0.00) | 0.1 (0.30)

15. Secondary Outcome: Number of Participants With Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categorization Mapped From Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS: a measure used to identify and assess participants at risk for suicide. It is a semi-structured interview that captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors. C-SSRS items were mapped to the following C-CASA categories: completed suicide, attempted suicide (actual attempt; aborted attempt; interrupted attempt), non-suicidal self-injurious behavior, preparatory acts, suicidal ideation (wish to be dead; non-specific active suicidal thoughts; active suicidal ideation with any methods [not plan], without intent to act; active suicidal ideation with some intent to act, without specific plan; active suicidal ideation with specific plan and intent; self-injurious behavior, no suicidal intent). C-CASA categories with at least 1 participant, for specified time points, for at least 1 reporting arm are reported below.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
Participants
  Week 6: Wish to be dead: number analyzed (Participants) | 6 | 11
  Week 6: Wish to be dead | 0 | 1
  Week 10: Wish to be dead: number analyzed (Participants) | 5 | 11
  Week 10: Wish to be dead | 0 | 1
  Week 26: Wish to be dead: number analyzed (Participants) | 8 | 13
  Week 26: Wish to be dead | 0 | 1
  Week 26: Non-specific Active Suicidal Thoughts: number analyzed (Participants) | 8 | 13
  Week 26: Non-specific Active Suicidal Thoughts | 0 | 1
  Week 26: Active Suicidal Thoughts With No Plan, Intent: number analyzed (Participants) | 8 | 13
  Week 26: Active Suicidal Thoughts With No Plan, Intent | 0 | 1

16. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale (CDRS-R) Total Score at Week 26
Description: CDRS-R: clinician-rated interview-based scale to assess 17 distinct symptom areas to derive an index of depression severity. Each symptom area was rated on a 7-point scale; range from 1 (no impairment) to 17 (maximum impairment). Total CDRS-R score was calculated as sum of responses for each 7 symptom areas. Total CDRS-R score ranged from 17 (no impairment) to 119 (maximum impairment); higher score indicated greater impairment.
Time Frame: Baseline (last measurement from A1281198), A1281201: Week 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Baseline | 68.2 (16.40) | 67.7 (13.28)
  Change at Week 26: number analyzed (Participants) | 8 | 11
  Change at Week 26 | 1.6 (11.60) | 7.2 (10.13)

17. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score at Week 1, 2, 6, 14, 22, 26
Description: YMRS: an 11-item scale that measured the severity of manic episodes. Four items (irritability, speech, thought content, and disruptive/ aggressive behavior) were rated on a scale from 0 (symptom absent) to 8 (symptom extremely severe). The remaining items were rated on a scale from 0 (symptom absent) to 4 (symptom extremely severe). YMRS total score was sum of score of all 11 items and ranged from 0 (no symptoms) to 60 (extreme severity of symptoms), higher score indicated higher severity of mania.
Time Frame: Baseline (last measurement from A1281198), A1281201: Week 1, 2, 6, 14, 22, 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Baseline | 12.7 (8.31) | 12.0 (5.46)
  Change at Week 1: number analyzed (Participants) | 9 | 12
  Change at Week 1 | 0.6 (10.71) | -5.5 (6.87)
  Change at Week 2: number analyzed (Participants) | 7 | 12
  Change at Week 2 | -3.1 (5.90) | -3.4 (7.42)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 1.3 (10.01) | -3.7 (7.71)
  Change at Week 14: number analyzed (Participants) | 5 | 11
  Change at Week 14 | 0.8 (8.84) | -5.8 (3.95)
  Change at Week 22: number analyzed (Participants) | 2 | 10
  Change at Week 22 | 0.5 (9.19) | -4.0 (7.29)
  Change at Week 26: number analyzed (Participants) | 8 | 13
  Change at Week 26 | -1.9 (4.85) | -6.4 (5.50)

18. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Week 1, 2, 4, 6, 10, 14, 18, 22, 26
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state. CGI-S score ranged from 1 (not ill at all) to 7 (among the most extremely ill), higher scores indicated more severity of illness.
Time Frame: Baseline (last measurement from A1281198), A1281201: Week 1, 2, 4, 6, 10, 14, 18, 22, 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Baseline | 2.7 (1.25) | 2.5 (0.97)
  Change at Week 1: number analyzed (Participants) | 9 | 12
  Change at Week 1 | 0.3 (1.12) | -0.3 (1.07)
  Chang at Week 2: number analyzed (Participants) | 7 | 12
  Chang at Week 2 | 0.1 (1.21) | -0.3 (0.98)
  Change at Week 4: number analyzed (Participants) | 7 | 12
  Change at Week 4 | 0.0 (1.00) | -0.2 (1.40)
  Change at Week 6: number analyzed (Participants) | 6 | 11
  Change at Week 6 | 0.5 (1.38) | 0.0 (1.26)
  Change at Week 10: number analyzed (Participants) | 5 | 11
  Change at Week 10 | -0.2 (0.84) | -0.1 (0.83)
  Change at Week 14: number analyzed (Participants) | 5 | 11
  Change at Week 14 | 0.0 (1.00) | -0.5 (1.04)
  Change at Week 18: number analyzed (Participants) | 3 | 11
  Change at Week 18 | -0.7 (1.15) | -0.4 (1.12)
  Change at Week 22: number analyzed (Participants) | 2 | 10
  Change at Week 22 | -1.0 (1.41) | -0.2 (1.14)
  Change at Week 26: number analyzed (Participants) | 8 | 13
  Change at Week 26 | -0.1 (1.25) | -0.5 (1.05)

19. Secondary Outcome: Change From Baseline in Children's Global Assessment Scale (CGAS) Total Score at Week 26
Description: CGAS: a clinician-rated global assessment item for children, based on symptoms and social functioning in home, school, and community settings. Scores ranged from 1 (extremely impaired) to 100 (doing very well), where higher levels indicate better health.
Time Frame: Baseline (last measurement from A1281198), A1281201: Week 26
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
Number analyzed (Participants) | 10 | 13
units on a scale
  Baseline | 68.2 (16.40) | 67.7 (13.28)
  Change at Week 26: number analyzed (Participants) | 8 | 11
  Change at Week 26 | 1.6 (11.60) | 7.2 (10.13)

ADVERSE EVENTS:
Time Frame: A1281201: Day 1 up to 35 days after last dose of study medication (maximum up to 31 Weeks)
Description: Same event may appear as both AE and SAE. An event may be categorized as serious in 1 participant and non-serious in other, or participant may experience both SAE and non-SAE. The safety analysis set included all participants who took at least 1 dose of study medication in this open-label extension study.
Arm/Group | Ziprasidone in A1281198 and A1281201 | Placebo in A1281198 Then Ziprasidone in A1281201
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/13
Other Adverse Events (participants affected / at risk) | 7/10 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone in A1281198 and A1281201 (N=10) | Placebo in A1281198 Then Ziprasidone in A1281201 (N=13)
Aggression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone in A1281198 and A1281201 (N=10) | Placebo in A1281198 Then Ziprasidone in A1281201 (N=13)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 7
Feeling abnormal (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Blood insulin increased (Investigations) | 1 | 0
Streptococcus test positive (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Akathisia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dystonia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 3 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures per study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT03768726/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/26/NCT03768726/SAP_001.pdf